CLINICAL TRIAL: NCT05296291
Title: RCT Study of Posterior Implant Supported Bridges Made of Various Prosthetic Materials
Brief Title: RCT: Titanium vs FCZ vs Zirconia Framework
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Branemarkkliniken (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1563
Record Dates: First submitted 2022-02-28; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Dental Prosthesis Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-translucent monolithic zirconia, (Active Comparator)
  Interventions: Device: High-translucent monolithic zirconia Bridge
- Zirconia ceramic with porcelain (Active Comparator)
  Interventions: Device: Zirconium oxide ceramics Framework
- Metal ceramics. (Active Comparator)
  Interventions: Device: Metal-ceramic Framework

INTERVENTIONS:
Device: High-translucent monolithic zirconia Bridge — Each patient will be treated according to standard of care with implants from Nobel Biocare, the Branmark system and then randomly assigned to receive a bridge made of either 1) metal ceramic (Nobel Procera, titanium skeleton), 2) zirconia ceramics (Nobel Procera zirconia skeleton) or 3) high-translucent monolithic zirconia (Nobel Procera).
  Arms: High-translucent monolithic zirconia,
Device: Zirconium oxide ceramics Framework — Each patient will be treated according to standard of care with implants from Nobel Biocare, the Branmark system and then randomly assigned to receive a bridge made of either 1) metal ceramic (Nobel Procera, titanium skeleton), 2) zirconia ceramics (Nobel Procera zirconia skeleton) or 3) high-translucent monolithic zirconia (Nobel Procera).
  Arms: Zirconia ceramic with porcelain
Device: Metal-ceramic Framework — Each patient will be treated according to standard of care with implants from Nobel Biocare, the Branmark system and then randomly assigned to receive a bridge made of either 1) metal ceramic (Nobel Procera, titanium skeleton), 2) zirconia ceramics (Nobel Procera zirconia skeleton) or 3) high-translucent monolithic zirconia (Nobel Procera).
  Arms: Metal ceramics.

SUMMARY:
In recent years, zirconia-based implant-supported bridge designs have begun to be used more and more as an alternative to metal ceramic bridges. Another new material that has been introduced in the clinic is the high translucent monolithic zirconia, which has only been investigated a few follow-up studies with short follow up duration.

The aim being to evaluate the clinical outcome of implant-anchored posterior bridges, made from

1. high-translucent monolithic zirconia,
2. zirconia ceramic with porcelain and
3. metal ceramics. The hypothesis is that high-translucent monolithic zirconia has lower rate of complications since surface porcelain veneering is not required.

A total of 60 research subjects will be included in the study. Patients in need of a permanent implant-supported bridge, located posterior of the canine in the upper or lower jaw will be asked for participation. Each subject will be treated according to standard treatment protocols with implants from Nobel Biocare, the Branemark implant system and then be randomly assigned to obtain one of the following three type of bridges.

20 research subjects will be included in each of the three study arms. The prosthetic treatment will be carried out according to standard clinic protocol.

All research subjects will be evaluated after 1, 3, 5 years. X-rays and photos will be taken at the installation of the bridges and after 1 and 5 years of follow-up or more frequent, depending on individual indication of the patient and the associated standard clinical care protocol.

Personal data, implant survival, marginal bone loss and biological and technical complications related to the implants will be recorded. Survival of the bridge, technical and biological complication related to the bridge will also be recorded

ELIGIBILITY:
Inclusion Criteria:

edentulous behind the canine in the maxilla or mandible

* older than 18 years

Exclusion Criteria:

* younger than 18 years
* active periodontitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complication rate | From placement of prosthetic Bridge until last follow-up of the study after 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- B R Å N E M A R K C L I N I C, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No